CLINICAL TRIAL: NCT04455425
Title: Descriptive Cohort of Acquired Syphlis by Non Sexual Contact
Brief Title: Acquired Syphlis by Non Sexual Contact
Status: Completed | Type: Observational
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Dr Jaime Altcheh, Principal Investigator, Hospital de Niños R. Gutierrez de Buenos Aires
Other Study IDs: Si non sexual
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Syphilis Acquired; Syphilis Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Syphilis is classically described as a sexually transmitted disease. As this source of contagious has been described long ago -mainly though by observation- when children presents with acquired syphilis, child abuse is always considered and must be ruled out by specialists in a careful evaluation.

However, muco-cutaneous lesions can be a contagious source for congenital syphilis; therefore the possibility of non-sexual transmission through intimate contact with infected people through humid lesions (such as in kisses, breastfeeding, food-handling) or contaminated fomites (towels, bed sheets, underwear, cups, pacifiers, cutlery) could be considered. Experts worldwide have observed this non-sexual transmission, as described in many reports in literature.

The investigators will study retrospectively patients from a cohort with non-sexual transmission. The diagnosis criteria used for acquired syphilis were as follows: age under 18 years with treponemic and nontreponemic positive tests, secondary-syphilis suspicious lesions and negative maternal syphilis serology. Nonsexual contagious was defined as contacts without physical and psychosocial indicators of sexual abuse according to current guides. In this cohort, in every case a psychosocial evaluation was completed with a written report in order to evaluate sexual contact probability.

The teamo will describe these patients clinical and laboratory findings, family and close acquaintances serologies and probable source of contagious.

ELIGIBILITY:
INCLUSION CRITERIA:

- Children with treponemic and non-treponemic positive tests with primary or secondary-syphilis suspicious lesions

EXCLUSION CRITERIA:

- Children with diagnose criteria positive for Congenital syphilis

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children from 0 to 18 years of age assisted at Parasitoloy and Chagas department from Children's Hospital in Buenos Aires, Argentina
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Describe diagnose process of a cohort of children with assumed non-sexual acquired syphilis | Past 20 years
  Describe the interdisciplinary approach of patients with acquired syphilis and how non-sexual transmission was assumed
Describe serology titers from patients with non - sexually acquired syphilis and from their close contacts | Past 20 years
  Investigators will report serology titers from patients with non - sexually acquired syphilis at diagnose and follow-up until cure, and from their close contacts at diagnose and during follow up of those resulting positive at contact screening
Describe reported symptoms and physical findings at diagnose and during follow-up f children with assumed non-sexual acquired syphilis and their close contacts | Past 20 years
  Investigators will describe symptoms and physical findings from patients with non - sexually acquired syphilis at diagnose and follow-up until cure, and from their close contacts at diagnose and during follow up of those resulting positive at contact screening

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Moscatelli, MD, Principal Investigator — Principal Investigator
Locations (1):
- Hospital de Niños Ricardo Gutierrez, Buenos Aires, Buenos Aires F.D., Argentina